CLINICAL TRIAL: NCT05345990
Title: Hepatitis B Immunoglobulins to Induce HBsAg Clearance in Patients With Chronic Hepatitis B (HBIG for Cure)
Brief Title: Treatment of Patients With Chronic Hepatitis B With Hepatitis B Immunoglobulins
Acronym: HBIG
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A full recruitment for the study was no longer expected.
Sponsor: Hannover Medical School (Other)
Collaborators: Biotest (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBIGforcure; 2021-005362-18 (EudraCT Number)
Record Dates: First submitted 2022-03-29; First posted 2022-04-26 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Chronic Hepatitis B
Keywords: Human hepatitis B Immunoglobulin
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — hepatitis B hyperimmune globulin

STUDY DESIGN:
Intervention Model Description: Patients treated in two cohorts for 12 weeks with hepatitis B immunoglobulins
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hepatitis B immunoglobulins (Experimental): 20 patients treated in two cohorts for 12 weeks with hepatitis B Immunoglobulins (HBIG, Hepatect®CP/ Zutectra®).
  Cohort A:
  10 HBsAg positive, HBeAg-negative patients being treated with anti-HBV nucleotide or nucleoside analogous (NAs) for at least 12 months before screening. HBV-DNA should be below the lower limit of detection at screening. HBsAg should be positive and below 100 IU/ml.
  Cohort B:
  10 HBsAg positive, HBeAg-negative patients untreated with NAs for at least 12 months before screening. Patients with HBV-DNA levels below 2000 IU/ml and ALT < 1.5 times upper the limit of normal. HBsAg should be positive and below 100 IU/ml.
  Trial duration: A recruiting period of approximately 6 months is planned. The total time per patient to complete all study visits is approximately 40 weeks including:
  * an 28 day screening period
  * an 12 week treatment period
  * an 24 week follow-up period
  Interventions: Drug: Human hepatitis B Immunoglobulin (Hepatect®CP/Zutectra®)

INTERVENTIONS:
Drug: Human hepatitis B Immunoglobulin (Hepatect®CP/Zutectra®) — Hepatect® is a solution to be administered Intravenously. Zutectra® is a solution to be administered subcutaneously.
  Treatment for 12 weeks with hepatitis B immunoglobulins with following administration scheme:
  D0: 10.000 IU Hepatect® i.v. D1-6: 500 IU Zutectra® s.c. D7: 10.000 IU Hepatect® i.v. D9- D84: 500 IU Zutectra® s.c. every 2nd day

SUMMARY:
This is an open-label, single arm (two cohorts), single-center, phase II pilot-study to provide preliminary evidence whether hepatitis B immunoglobulins (HBIG) are efficacious and can be safely used in patients with chronic Hepatitis B Virus (HBV) infection.

A total of 20 patients (male or female adults aged ≥ 18 years) will be enrolled in the study and receive hepatitis B immunoglobulins Hepatect®CP and Zutectra®.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study:

1. Willing and able to provide written informed consent
2. Male or female, age ≥ 18 years
3. Confirmation of chronic HBV infection documented by:

   positive HBsAg at least 12 months before screening
4. Cohort A: NA treatment for at least 12 months before screening. HBV-DNA should be below the lower limit of detection at screening. HBsAg positive and <100 IU/ml. HBeAg negative.
5. Cohort B: Untreated with NAs for at least 12 months before screening. HBV-DNA < 2000 IU/ml. HBsAg positive and < 100 IU/ml. HBeAg-negative.
6. Subject has not been treated with any investigational drug or device within 42 days before the screening visit or within 5 half-lives for investigational drugs, whichever is longer.
7. Transient Elastography (FibroScan) < 7.5 kPa at screening.
8. ALT levels < 1.5 times of upper the limit of normal at screening for both cohorts
9. Body mass idex (BMI) > 18kg/m²
10. A negative serum pregnancy test is required for female subjects (unless surgically sterile or women > 54 years of age with cessation for > 24 months of previously occurring menses). Complete abstinence from intercourse. Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) is not permitted. Or Consistent and correct use of 1 of the following methods of birth control listed below, in addition to a male partner who correctly uses a condom, from the date of Screening until the end of FU:

    * intrauterine device (IUD) with a failure rate of < 1% per year
    * bilateral tubal sterilization
    * vasectomy in male partner
    * hormone-containing contraceptive:

      * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

        * oral
        * intravaginal
        * transdermal
      * progestogen-only hormonal contraception associated with inhibition of ovulation:

        * oral
        * injectable
        * implantable
11. Subject must be able to comply with the dosing instructions for study drug administration and be able to complete the study schedule of assessments

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria are not to be enrolled in this study:

1. Clinically significant illness (other than hepatitis B) or any other major medical disorder that, in the opinion of the investigator, may interfere with subject treatment, assessment or compliance with the protocol. Subjects currently under evaluation for a potentially clinically significant illness (other than hepatitis B) are also excluded.
2. Co-infection with hepatitis C virus (defined as HCV RNA positive. HCV RNA negative/anti-HCV-positive patients can be included) or co-infection with HIV.
3. Clinical hepatic decompensation (i.e. clinical ascites, encephalopathy or variceal hemorrhage).
4. Psychiatric hospitalization, suicide attempt, and/or a period of disability as a result of their psychiatric illness within the last 2 years. Subjects with psychiatric illness that is well-controlled on a stable treatment regimen for at least 12 months prior to screening or has not required medication in the last 12 months may be included.
5. Significant drug allergy (such as anaphylaxis or hepatotoxicity).
6. Pregnant or nursing female or male with pregnant female partner
7. Clinically relevant drug or alcohol abuse within 12 months of screening including any uncontrolled drug use within 6 months of screening. A positive drug screen will exclude subjects unless it can be explained by a prescribed medication. The investigator must approve medication, the diagnosis and prescription. Uncontrolled users of intravenous drugs will not be permitted to enroll in the study.
8. live-attenuated virus vaccinations such as: measles, mumps, rubella and varicella 4 weeks before and up to three months after administration of hepatitis B immunoglobulins. If not required by an emergency situation, passive or active immunizations or administration of plasma preparations or of other immunoglobulins is not allowed during the study
9. A recent SARS-COV2 infection in the last 4 weeks prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of 12-weeks treatment with hepatitis B immunoglobulins in two different cohorts of patients with chronic hepatitis B defined by the proportion of subjects being HBsAg negative at treatment week 12 | week 12 of antiviral therapy
  Primary efficiency endpoint: HBsAg negativity at week 12 of antiviral therapy

SECONDARY OUTCOMES:
To analyze the change/decline of HBsAg during treatment | week 1, 2, 4, 8 and 12 of treatment
  Secondary endpoint: HBsAg change/decline at weeks 1, 2, 4, 8 and 12 of treatment
To evaluate the post-treatment HBsAg kinetics/response | Follow-up (FU) week 2, FU week 4, FU week 12 and FU week 24
  Secondary endpoint: Post-treatment HBsAg negativity up to FU week 24
To determine HBV-DNA levels during and after treatment with hepatitis B immunoglobulins | screening, day 0, day 1, day 3, day 7, day 28, day 42, day 84, FU week 12 and FU week 24
  Secondary endpoint: HBV DNA levels during and after hepatitis B immunoglobulin treatment will be reported for each cohort.
To evaluate the biochemical disease activity (normalization of serum ALT levels) | week 12 of treatment
  Secondary endpoint: biochemical response (proportion of subjects who reached ALT normalization (ALT ≤ ULN) at week 12 of treatment)
To determine the quality of life by SF-36 questionnaire | day 0, day 84, FU week 12, FU week 24
  Secondary endpoint: quality of life during treatment and follow-up (SF-36)
Assessment of safety by collection of adverse events (AEs) as frequencies (absolute/relative). | day 0, day 1, day 3, day 7, day 14, day 21, day 28, day 42, day 56, day 84, FU week 2, FU week 4, FU week 12, FU week 24
  Adverse events (AEs) will be collected throughout the study (upon first administration of the IMPs up to 24 weeks after discontinuation of therapy, FU24) and will be reported with absolute and relative frequencies along with the corresponding 95% confidence intervals

CONTACTS AND LOCATIONS:
Overall Officials: Heiner Wedemeyer, Prof., Principal Investigator — Hannover Medical School, Department of Gastroenterology, Hepatology and Endocrinology
Locations (1):
- Hannover Medical School, Department for Gastroenterology, Hepatology and Endocrinology, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No